CLINICAL TRIAL: NCT00934830
Title: Antibiotics Versus Therapeutic Ultrasound for Treatment of Sinusitis: a Randomized Clinical Trial
Brief Title: Antibiotics Versus Therapeutic Ultrasound for Sinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sør-Trøndelag chapter of the Norwegian Physiotherapist Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELI-107-04(REK)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Sinusitis
Keywords: Antibiotic; Ultrasound; Efficacy; Treatment
MeSH Terms: conditions — Sinusitis | interventions — Anti-Bacterial Agents; Amoxicillin; Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic (Active Comparator)
  Interventions: Drug: Antibiotic (Amoxicillin)
- Therapeutic ultrasound (Experimental)
  Interventions: Other: Therapeutic ultrasound

INTERVENTIONS:
Drug: Antibiotic (Amoxicillin) — 500 mg, 3 times per day for 10 days
  Arms: Antibiotic
Other: Therapeutic ultrasound — 1.0 W/cm2 in continuous mode for 10 minutes once a day for 4 consecutive days.
  Arms: Therapeutic ultrasound

SUMMARY:
Question: Is the effect of therapeutic ultrasound equally effective to antibiotic for treatment of sinusitis? Design: A randomized clinical trial with concealed allocation, self-assessment by the subjects and intention-to-treat analysis.

DETAILED DESCRIPTION:
Subjects (n=48) with clinically diagnosed acute bacterial rhinosinusitis (ABRS)will included. The antibiotic group will receive amoxicillin (500 mg) 3 times per day for 10 days. The ultrasound group will receive therapeutic ultrasound over sinuses at 1.0 W/cm2 in continuous mode for 10 minutes once a day for 4 consecutive days. Improvement of symptoms (pain and congestion; numeric rating scale; 0-10) from day 1 to days 4 and 21 will be recorded. Relapses, side-effects and satisfaction with treatment will be assessed at one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Pain when bending forward, headache, pain in the teeth, purulent nasal secretion, "double worsening" and white blood cell count (WBC).
* Patients eligible for the study had to meet one of the first three criteria (pain when bending forward, headache, pain in the teeth) and all of the other indicators (purulent nasal secretion, double worsening, a left handed displacement of lymphocytes and a right handed displacement of granulocytes on the WBC as indication of bacterial infection).
* Subjects over 15 years of age were included.

Exclusion Criteria:

* Subjects with any kind of antibiotic or allergic treatment within the last three weeks.
* Antibiotic intolerance.
* Pregnant women.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pain and congestion over in forehead, around nose and pain in the teeth | Day 1, 4 and 21, and one-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ottar Vasseljen, PhD, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Røros Medical Center, Røros, Norway

REFERENCES:
- [Result] Hosoien E, Lund AB, Vasseljen O. Similar effect of therapeutic ultrasound and antibiotics for acute bacterial rhinosinusitis: a randomised trial. J Physiother. 2010;56(1):29-32. PMID 20500134